CLINICAL TRIAL: NCT02467413
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel, Phase II Study to Evaluate Efficacy and Safety of BAC in Patient With Alzheimer's Disease or Vascular Dementia
Brief Title: BAC in Patient With Alzheimer's Disease or Vascular Dementia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn before participants were enrolled.
Sponsor: Charsire Biotechnology Corp. (Industry)
Collaborators: A2 Healthcare Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAC-01
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Alzheimer's Disease; Vascular Dementia
Keywords: Alzheimer's Disease; Vascular Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BAC treatment group (Active Comparator): BAC, topical application on external nasal skin, scalp, and neck, 30g/day, 2 times daily, for 12 weeks
  Interventions: Drug: BAC
- BAC Matched vehicle (Placebo Comparator): BAC Matched vehicle, topical application on external nasal skin, scalp, and neck, 30g/day, 2 times daily, for 12 weeks
  Interventions: Other: BAC Matched Vehicle

INTERVENTIONS:
Drug: BAC — (vapor fraction from seeds of Glycine max (L.) Merr. and composition thereof)
  Other Names: CSTC1-BAC
  Arms: BAC treatment group
Other: BAC Matched Vehicle — BAC Matched Vehicle
  Arms: BAC Matched vehicle

SUMMARY:
The primary objective of this study is to evaluate the efficacy of BAC patients with Alzheimer's disease or vascular dementia.The secondary objective of this study is to evaluate the safety of BAC patients with Alzheimer's disease or vascular dementia.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, vehicle-controlled and parallel trial to evaluate the efficacy and safety of BAC in patients with Alzheimer's disease or vascular dementia. The investigation product, BAC, is a potential anti-inflammatory agent consisted of Multi-Glycan Complex (MGC) from the Soybean extract. It aims to reduce the neruoinflammation in the Alzhemimer's disease and vascular dementia.

Eligible patients will be randomly assigned to receive either one of topical application of BAC or BAC matched vehicle, topical application on external nasal skin, scalp, and neck, 30mL/day, 2 times daily.

The treatment duration for each patient is 12 weeks, which consists of 6 visits located at Screening, Baseline (Week 0), Weeks -2, -4, -8, and -12. During the treatment period, patients may continue to receive routinely used medications or treatments for Alzheimer's disease or vascular dementia except those prohibited under this protocol.

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible for the study if all of the following apply:

1. With either gender aged at least 40 years old
2. With a diagnosis of one of the following disease i. Vascular dementia according to the NINDS-AIREN International Workshop criteria or ii. Alzheimer's disease according to the NIAAA criteria iii. "Mixed" dementia (possible Alzheimer's disease with cerebrovascular disease) according to the NIAAA criteria

   Note:
   1. NINDS-AIREN: National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherche et l'Enseignement en Neurosciences
   2. NIAAA: National Institute on Aging-Alzheimer's Association
3. With mild-to-moderate dementia (score of the Mini-Mental State Examination (MMSE) defined as between 10 to 24)
4. Able to read, write, communicate, and understand cognitive testing instructions
5. Having a responsible caregiver who spends adequate time daily with the patient; the caregiver will accompany the patient to all clinic visits during the study and supervise all study dosing requirements and concomitant medications
6. Signed, by patients and the responsible caregiver, the written informed consent form

Exclusion Criteria:

1. With large-artery stroke (thrombotic stroke)
2. With radiological evidence of other brain disorders (subdural hematoma, post-traumatic / post-surgery)
3. With dementia caused by other brain diseases except Alzheimer's disease and vascular dementia (e.g. Parkinson's disease, demyelinated disease of the central nervous system, tumor, hydrocephalus, head injury, central nervous system infection including syphilis, acquired immune deficiency syndrome, etc.)
4. With clinical evidence of pulmonary, hepatic, gastrointestinal, metabolic, endocrine or other life threatening diseases judged by investigators not suitable to enter the study
5. With clinically unstable hypertension, diabetes mellitus, and cardiac disease for the last 3 months
6. With history of stroke and hospitalized for stroke in the previous 3 months
7. With history of alcohol or drug abuse
8. With one of the following abnormal laboratory parameters: hemoglobin < 10 mg/dL or platelet < 100*109/L; creatinine or total bilirubin more than 1.5 times the upper limit value; alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphates (ALP), or γ-glutamyl transferase (γ-GT) more than 2 times the upper limit of normal
9. With depression, not well-controlled with medications.
10. With any uncontrolled illness judged by the investigator that entering the trial may be detrimental to the patient
11. With known or suspected hypersensitivity to any ingredients of study product and vehicle
12. Pregnant or lactating or premenopausal with childbearing potential but not taking reliable contraceptive method(s) during the study period
13. Enrollment in any investigational drug trial within 4 weeks before entering this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-30 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale- Cognitive (ADAS-cog) score at Week-12 visit compared to baseline | Weeks 12
  The Alzheimer's Disease Assessment Scale- Cognitive (ADAS-Cog) Subscale test is the standard assessment tool and one of the most popular cognitive testing instrument in clinical trials.

SECONDARY OUTCOMES:
Change in ADAS-cog score at all post treatment visits (except Week-12 visit) compared to baseline | Weeks 4, 8, 12
  The Alzheimer's Disease Assessment Scale- Cognitive (ADAS-Cog) Subscale test is the standard assessment tool and one of the most popular cognitive testing instrument in clinical trials.
Clinician's Interview Based Impression of Change-Plus Caregiver Input (CIBIC-plus) score at all post treatment visits | Weeks 4, 8, 12
  This is a global measure of detectable change in cognition, function and behavior.
Change in Activities of Daily Living (ADL) score at all post treatment visits compared to baseline | Weeks 4, 8, 12
  An inventory of informant based items to assess activities of daily living and instrumental activities of daily living, i.e. functional performance, of Alzheimer's disease (AD).
Change in Mini-Mental State Examination (MMSE) score at all post treatment visits compared to baseline | Weeks 4, 8, 12
  This is a multi-item instrument that examines orientation, registration, attention, calculation, recall, visuospatial abilities and language. The score ranges from 0 to 30, with higher scores indicating better cognitive function. MMSE was measured at Screening, Randomization/Baseline, Week 4, Week 8, and Week 12.
Change in Neuropsychiatric Inventory (NPI) score at all post treatment visits compared to baseline | Weeks 4, 8, 12
  The NPI is the behavior instrument most widely used in clinical trials of anti-dementia agents. The NPI uses a screening strategy to minimize administration time, examining and scoring only those behavioral domains with positive responses to screening questions. Both the frequency and the severity of each behavior are determined. Information for the NPI is obtained from a caregiver familiar with the patient's behavior. The NPI assesses 12 behavioral domains (12-item NPI) common in dementia. Each NPI domain is scored by the caregiver based on a standardized interview administered by the clinician. NPI-12 Caregiver Distress score is scored for associated caregiver distress from 0 (no distress) to 5 (very severe or extreme). Higher scores indicate greater distress. NPI was measured at Randomization/Baseline, Week 4, Week 8, and Week 12.
Adverse event incidence | Baseline, Weeks 4, 8, 12
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a study medication and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a study medication, whether or not related to the study medication. Laboratory abnormalities should not be recorded as AEs unless determined to be clinically significant by the Investigator. The number of participants with adverse events within the BAC and placebo groups was determined.
Change in physical examination results | Weeks 4, 8, 12
  Items include general appearance, skin, eyes, ears, nose, throat, head and neck, heart, joints, chest and lungs, abdomen, lymph nodes, musculoskeletal, nervous system, and others.
Net change from baseline in laboratory test results | Weeks 4, 8, 12
  Items include blood pressures, pulse rate, respiratory rate, and body temperature.
Net change from baseline in vital signs | Weeks 4, 8, 12]
  Items include 1. hematology: hemoglobin, hematocrit, red blood cell (RBC), platelet, white blood cell (WBC) with differential counts; 2. Biochemistry: aspartate aminotransferase (AST), alanine aminotransferase (ALT), γ-glutamyl transferase (γ-GT), serum creatinine, blood urea nitrogen (BUN), albumin, total protein, alkaline phosphatase, total bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Pai Ming-Chyi, PhD, Principal Investigator — Neurology National Cheng Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan